CLINICAL TRIAL: NCT05654454
Title: Randomized Double Blind Phase III Trial Comparing Safety and Efficacy of Bevacizumab (Mabscale LLC, Russia) + Paclitaxel + Carboplatin to Avastin® + Paclitaxel + Carboplatin in Inoperable or Advanced Non-squamous Non-small-cell Lung Cancer
Brief Title: A Safety and Efficacy Study of Bevacizumab, Paclitaxel, Carboplatin Compared to Avastin® in Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mabscale, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BEV-III/2022
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bevacizumab with Paclitaxel and Carboplatin (Experimental): Patients will begin Period 1 receiving bevacizumab combination therapy (Bevacizumab 15 mg/kg IV + Paclitaxel 175 mg/m2 + IV Carboplatin AUC 6 IV) on Day 0 of Cycle 1 for up to 6 cycles of therapy. Each cycle will consist of 3 weeks (21 days ± 3 days) and a cycle will start with the administration of bevacizumab (produced by Mabscale, LLC).
  In Period 2, eligible patients will continue to receive bevacizumab (produced by Mabscale, LLC) every 3 weeks as monotherapy.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin
- Avastin® with Paclitaxel and Carboplatin (Active Comparator): Patients will begin Period 1 receiving bevacizumab combination therapy ( Avastin® 15 mg/kg IV + Paclitaxel 175 mg/m2 IV + Carboplatin AUC 6 IV) on Day 0 of Cycle 1 for up to 6 cycles of therapy. Each cycle will consist of 3 weeks (21 days ± 3 days) and a cycle will start with the administration of bevacizumab (as Avastin®).
  In Period 2, eligible patients will continue to receive bevacizumab (Avastin®) every 3 weeks as monotherapy.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 15 mg/kg
Drug: Paclitaxel — Paclitaxel 175 mg/m2
Drug: Carboplatin — Carboplatin AUC 6

SUMMARY:
BEV-III/2022 is a double-blind randomized multicenter clinical trial comparing efficacy of bevacizumab (manufactured by Mabscale, LLC) and paclitaxel plus carboplatin to Avastin® and paclitaxel plus carboplatin in first-line treatment for patients with advanced (unresectable, locally advanced, recurrent or metastatic) non-squamous NSCLC. The purpose of the study is to demonstrate equivalence of efficacy and safety of bevacizumab (manufactured by Mabscale, LLC) to Avastin®. Study includes pharmacokinetics assessment.

DETAILED DESCRIPTION:
Bevacizumab is a monoclonal antibody currently being developed by Mabscale LLC, as a proposed biosimilar to Avastin®, which is approved as first line treatment in combination with carboplatin and paclitaxel for patients with unresectable, locally advanced, recurrent or metastatic non-squamous Non-Small Cell Lung Cancer. This randomized equivalence study is designed to meet the regulatory requirement for approval of a biosimilar product.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male and female patients at least 18 years of age
* Newly diagnosed Stage IIIB/C or IV non-small cell lung cancer (according to Revised Cancer Staging by American Joint Committee on Cancer (AJCC) and the International Union Against Cancer (UICC) 8th edition) or recurrent non-small cell lung cancer (NSCLC)
* Histologically or cytologically confirmed diagnosis of predominately non-squamous NSCLC
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Be eligible to receive study treatment of bevacizumab, paclitaxel, and carboplatin based on local standard of care, for the treatment of advanced or metastatic non-squamous NSCLC
* Presence of at least 1 measurable tumour as defined by modified Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
* Neutrophils ≥ 1,5 × 10^9/L
* Platelets ≥ 100 × 10^9/L
* Haemoglobin ≥ 90 g/L
* Bilirubin level ≤ 1.5 × upper limit of normal (ULN)
* Aspartate-aminotransferase (AST) and alanine-aminotransferase (ALT) levels < 3 × ULN (< 5 × ULN for patients with liver metastases)
* Alkaline phosphatase level < 3 × ULN (< 5 × ULN for patients with liver or bone metastases)

Exclusion Criteria:

* Known sensitizing EGFR mutations or ALK translocation positive mutations
* Evidence of a tumor that compresses or invades major blood vessels or tumor cavitation that is likely to bleed
* Major surgery 28 days before inclusion into the study
* Minor surgery 7 days before inclusion into the study
* Stage II or higher of neuropathy or ototoxicity according to Common Terminology Criteria for Adverse Events (CTCAE) v.5.0, excluding trauma
* Life expectancy less than 6 months
* Metastases to central nervous system or carcinomatous meningitis
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) at Week 18 | 18 weeks from randomisation
  Objective response rate was assigned for a subject if the subject displayed either complete response (CR) or partial response (PR) per RECIST version 1.1 at Week 18, as assessed by independent radiological review committee (IRC).

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | At week 18 and 42 from randomisation
  Progression-free survival was defined as the time from randomization to subsequent confirmed progression per RECIST version 1.1, or death (whichever occurred first), measured in weeks and months. For PFS assessment clinical progression (i.e., treatment discontinuation due to progression of disease) was also considered as an event.
Overall Survival (OS) | At week 18 and 42 from randomisation
  Overall survival was defined as the time from randomization to subsequent death, measured in weeks and months.
Duration of response (DOR) | 48 weeks
  Duration of responce was defined as the time from responce to treatment till progression or death.

CONTACTS AND LOCATIONS:
Locations (28):
- Russia (28):
  - Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk
  - State Budget Healthcare Institution Ivanovo Regional Oncology Dispensary, Ivanovo
  - Kaluga Regional Clinical Oncology Dispensary, Kaluga
  - Regional clinical oncological dispensary n.a.Sigal, Kazan'
  - Burdenko Main Military Clinical Hospital, Moscow
  - Hadassah Medical Moscow, Moscow
  - National Medical Oncology Research Center n.a. N.N. Blokhina, Moscow
  - Murmansk Regional Clinical Hospital, Murmansk
  - Nizhny Novgorod Regional Oncology Dispensary, Nizhny Novgorod
  - Novosibirsk oncologic dispensary, Novosibirsk
  - Omsk clinical oncologic dispensary, Omsk
  - Perm Edge Clinical Hospital, Perm
  - Perm Regional Clinical Hospital, Perm
  - Euromedservice medical center, Pushkin
  - Clinical Hospital RZD-Medicine, Saint Petersburg
  - Euro Cityclinic, Saint Petersburg
  - Leningrad regional clinical hospital (prev.Oncological dispensary n.a.Roman), Saint Petersburg
  - Leningrad regional clinical hospital, Saint Petersburg
  - National Medical Research Center of Oncology N.A. N.N. Petrov, Saint Petersburg
  - Northwestern Center for Evidence-Based Medicine, Saint Petersburg
  - Medical University "Reaviz", Samara
  - Smolensk oncologic dispensary, Smolensk
  - Smolensk Regional Clinical Hospital, Smolensk
  - Tverskoy Regional Oncological Dispensary, Tver'
  - Bashkir State Medical University, Ufa
  - Oblastnoy Clinical Oncological Dispansery, Veliky Novgorod
  - Volgograd Regional Clinical Oncology Dispensary, Volgograd
  - Regional Clinical Oncological Hospital, Yaroslavl